CLINICAL TRIAL: NCT03525392
Title: An International Multicentre, Open-Label First in Human Phase I/II Study to Evaluate the Safety, Tolerability, Biodistribution and Antitumour Activity of 177Lu-3BP-227 for the Treatment of Subjects With Solid Tumours Expressing Neurotensin Receptor 1
Brief Title: Study to Evaluate the Safety and Activity (Including Distribution) of 177Lu-3BP-227 in Subjects With Solid Tumours Expressing Neurotensin Receptor Type 1.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to agreement to transfer rights for IPN01087 to an external partner, not due to safety concerns
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-FR-01087-001; 2017-001263-20 (EudraCT Number)
Record Dates: First submitted 2018-05-03; First posted 2018-05-15 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Colorectal Cancer; Gastric Cancer; Squamous Cell Carcinoma of the Head and Neck; Bone Cancer; Advanced Cancer; Recurrent Disease; Metastatic Tumours
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Bone Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-3BP-227 (Experimental): Screening: 177Lu-IPN01087 - 25 µg 3BP-227 (IPN01087) per 1 GBq of 177Lu. 1 GBq in a total volume of 10 mL.
  Treatment phase: 177Lu-IPN01087 - 2.5 to 7.5 GBq escalation dose of 177Lu-3BP-227 (IPN01087) in a total volume of 20 mL for each cycle of administration (2 cycles plus 4 optional additional).
  Interventions: Drug: 177Lu-3BP-227 (also called 177Lu-IPN01087)

INTERVENTIONS:
Drug: 177Lu-3BP-227 (also called 177Lu-IPN01087) — The cumulative activity of the treatment investigational medicinal product (IMP) formulation will be administered in two intravenous (i.v.) infusions separated by at least 4 weeks (28 days). Up to 6 administrations can be given (2 cycles plus 4 optional additional)
  Other Names: 177Lu-IPN01087

SUMMARY:
This study was conducted to advance new treatment for patients with metastatic or locally advanced cancers expressing Neurotensin receptor 1 (NTSR1). This study was the first time the investigational drug called 177Lu-3BP-227 was administered to patients under controlled conditions of a clinical study.

The purpose of this study was to evaluate how safe the investigational drug is as well to verify how well it is tolerated by patients after several intravenous administrations. In addition, the effect of the study drug on tumoral lesions and how it distributes throughout the body and at which rate it is removed from the body was evaluated. Since 177Lu-3BP-227 is a radio-labelled drug, it also measured how the emitted radiation is distributed throughout the body (dosimetry).

The study consisted of a phase I dose escalation part. The study originally planned to include a phase II study however due to early termination (not due to safety concerns) the study did not progress to phase II and was stopped during phase I. For the phase I dose escalation part, it was anticipated that approximately 30 subjects will be included, in up to six escalation steps. No expansion cohorts were implemented.

ELIGIBILITY:
Inclusion Criteria :

* Signed informed consent form prior to all study procedures
* Aged 18 years or older.
* Histologically or cytologically confirmed unresectable locally advanced or metastatic disease and has received prior lines of standard-of-care chemotherapy/treatment and has no further suitable treatment options and documented decision by a multidisciplinary oncology board including a specialist of the concerned pathology.
* Subjects have (a) pancreatic ductal adenocarcinoma (PDAC), or (b) colorectal adenocarcinoma (CRC), or (c) gastric adenocarcinoma (GC), or (d) gastrointestinal stromal tumours (GIST), or (e) squamous-cell carcinoma of head and neck (SCCHN), or (f) Ewing Sarcoma (ES)
* Tumour showing: (a) by uptake of 177Lu-3BP-227 (screening formulation) in known primary or metastatic sites as judged by the investigator to be greater than background; or (b) uptake of 111In 3BP 227 in known primary or metastatic sites (for subjects who participated in Study D FR 01087 002) as judged by the investigator to be greater than background.
* Measurable disease (based on RECIST version1.1).
* Documentation of progressive disease in the 6 months prior to study start (treatment).
* Eastern Cooperative Oncology Group performance status of 0 or 1 (unless if disability is related to surgery in ES and Agreed with the Sponsor).
* Adequate organ function as evidenced by: (a) Leukocytes ≥3000/μL (b) Absolute neutrophil count ≥1500/µL (c) Platelets ≥75,000/µL (d) Hb >9 g/dL or >10 g/dL (if history of cardiac disease) (e) Total serum bilirubin ≤2 times upper normal institutional limits (ULN) (f) Aspartate aminotransferase/alanine aminotransferase (ALT) ≤2.5×ULN (or ≤5×ULN, if subject has liver metastases) (g) Estimated glomerular filtration rate (eGFR) ≥55 mL/min.
* Estimated life expectancy >3 months.
* Female subjects must not be pregnant or lactating at study entry and during the course of the study and must not become pregnant for at least 6 months following the last study treatment. Women of childbearing potential must agree to use a highly effective method of contraception
* For male subjects, must not father children during the study and for at least 6 months after the last study treatment and in addition must agree to use a condom for this period to protect his partner from contamination with the IMP. For males with partners who are of child bearing potential, effective contraception is a combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier methods), but these are not considered to be highly effective. A man is considered to be infertile if he has had bilateral orchidectomy or successful vasectomy. Effective contraception includes a female partner of childbearing potential if she is using highly efficacious contraception, but the male subject must agree to use a condom to protect his partner as described above.
* Must be willing and able to comply with study restrictions and to remain at the clinic for the required time during the study period and willing to return to the clinic for the follow-up evaluation, as specified in the protocol.

Exclusion Criteria :

* Prior treatment received (a) Any antitumor treatment since last documented disease progression (b) Any chemotherapy within 3 weeks or nitrosourea within 6 weeks prior to first treatment investigational medicinal product (IMP) administration (c) Any curative radiotherapy within 4 weeks, or palliative radiotherapy within 7 days prior to first treatment IMP administration (d) Any monoclonal antibodies within 4 weeks or tyrosine kinases inhibitors within 2 weeks prior to the first treatment IMP administration, (e) Any other IMP within 2 weeks prior to first treatment IMP administration, if the previous compound is a mechanism-based molecularly targeted agent whose half-life (t1/2) is not well-characterized.
* Brain metastases.
* Nephrectomy, renal transplant or concomitant nephrotoxic therapy putting the subject at high risk of renal toxicity during the study.
* Only non-measurable metastatic bone lesions
* Existing or planned colostomy during study participation.
* Any history of inflammatory bowel disease.
* Any uncontrolled significant medical, psychiatric or surgical condition or laboratory finding, that would pose a risk to subject safety or interfere with study participation or interpretation of individual subject results.
* Clinically significant abnormalities on electrocardiogram (ECG) at screening including corrected QT interval (Fridericia's formula) >450 msec for males or 470 msec for females at screening.
* Previously received external beam irradiation to a field that includes more than 30% of the bone marrow or kidneys.
* Any unresolved NCI-CTCAE Grade 2 or higher toxicity (except alopecia) from previous antitumor treatment and/or medical/surgical procedures/interventions.
* Known allergy to IMP or its excipients administered in this study, including imaging contrast media.
* Positive pregnancy test (female subjects).
* Likely to be uncompliant or uncooperative during the study, in the judgment of the investigator.
* Unable to understand the nature, scope, and possible consequences of the study, in the judgment of the investigator.
* Sponsor employees or investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Institut Jules Bordet, Brussels, Belgium
- France (3):
  - Centre Léon Bérard, Lyon
  - CHU Timone, Marseille
  - CHU Hôtel Dieu, Nantes
- University Medical Center Groningen, Groningen, Netherlands
- Switzerland (2):
  - CHU Vaudois, Lausanne
  - Universitäts Spital Zürich, Zurich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1/2 first in human study was conducted in participants with unresectable, locally advanced or metastatic solid tumors expressing neurotensin receptor 1 (NTSR1) at 9 investigational sites in Belgium, France, the Netherlands, Switzerland and USA between 03 May 2018 and 28 April 2021. The sponsor terminated the study early during Cohort 5 in phase 1 dose escalation; phase 1 dose expansion and phase 2 were not started.
Pre-assignment Details: For phase 1, the core trial was up to 19 weeks (including screening) and comprised of 2 treatment cycles. If a participant had clinical benefit (Investigator judgment), they could receive up to 4 additional cycles after end of core trial (EOCT) provided certain other criteria were met. Long-term follow-up period was up to 5 years. Due to early termination, only results of the core trial are presented. 14 participants received a therapeutic dose of 177Lu-3BP-227 in phase 1 of the study.
Groups:
- Cohort 1: 177Lu-3BP-227 2.5 GBq: Participants received 177Lu-3BP-227 2.5 Gigabecquerel (GBq) fractionated into 2 intravenous (IV) administrations separated by 4 to 5 weeks during the core trial period.
- Cohort 2: 177Lu-3BP-227 4.0 GBq: Participants received 177Lu-3BP-227 4.0 GBq fractionated into 2 IV administrations separated by 4 to 5 weeks during the core trial period.
- Cohort 3: 177Lu-3BP-227 5.5 GBq: Participants received 177Lu-3BP-227 5.5 GBq fractionated into 2 IV administrations separated by 4 to 5 weeks during the core trial period.
- Cohort 4: 177Lu-3BP-227 6.5 GBq: Participants received 177Lu-3BP-227 6.5 GBq fractionated into 2 IV administrations separated by 4 to 5 weeks during the core trial period.
- Cohort 5: 177Lu-3BP-227 7.5 GBq: Participants received 177Lu-3BP-227 7.5 GBq fractionated into 2 IV administrations separated by 4 to 5 weeks during the core trial period.
Period: Overall Study
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Started | 2 | 3 | 5 | 3 | 1
Completed (Completed the EOCT.) | 1 | 2 | 2 | 0 | 0
Not Completed | 1 | 1 | 3 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Included population contained all screened participants who were included in the study and received the therapeutic dose.
Groups:
- Cohort 1: 177Lu-3BP-227 2.5 GBq: Participants received 177Lu-3BP-227 2.5 GBq fractionated into 2 IV administrations separated by 4 to 5 weeks during the core trial period.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq | Total
Number analyzed (Participants) | 2 | 3 | 5 | 3 | 1 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (4.2) | 64.3 (16.2) | 64.0 (7.2) | 66.3 (9.1) | 77.0 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 66.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 0 | 4
  Male | 2 | 2 | 4 | 1 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Not Collected | 2 | 3 | 5 | 0 | 0 | 10
  White | 0 | 0 | 0 | 3 | 1 | 4
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black / African American | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian / Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  American Indian / Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5 | 3 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLTs were defined for a list of predefined study medication-related adverse events (AEs) as specified in the protocol, according to the National Cancer Institute - Common Terminology Criteria for Adverse Events scale version 5.0 that occurred during the defined DLT assessment period (during Cycle 1 or 2).
Time Frame: From the start of the first study medication (Cycle 1 Day 1) up to EOCT, maximum of 16 weeks.
Population: Safety population contained all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Number analyzed (Participants) | 2 | 3 | 5 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Phase 1: Maximum Uptake (%) of 177Lu-3BP-227 at Target Lesions and Discernible Organs
Description: 177Lu-3BP-227 uptake in organs and lesions was evaluated centrally, using nuclear medicine images, as part of the dosimetry workflow. Uptake activity for organs of interest (i.e., body, bone marrow, left kidney, right kidney, healthy liver, and spleen) was determined. The uptake activity was expressed relatively to the injected 177Lu-3BP-227 activity calculated as the ratio of the uptake activity divided by the administered activity at the time of injection.
Time Frame: Measurements were performed at 0 to 1 hours, 2 to 4 hours, 16 to 24 hours, 40 to 48 hours, 72 to 96 hours post infusion in each treatment cycle.
Population: Dosimetry population included all participants with organ dosimetry data and with no major protocol deviations with an impact on dosimetry analysis. Since the study drug administered to different groups had same composition/specific activity, no difference in drug distribution was expected between groups. Because uptake results were expressed as percentage of administered 177Lu-3BP-227 activity, no difference in uptake was expected between groups and results were reported combining all groups.
Measure: Median (Full Range); unit: percentage of injected 177Lu-3BP-227
Units Other Than Participants: Observations
Groups:
- All Participants: Participants received 177Lu-3BP-227 dose range of 2.5 to 7.5 GBq fractionated into 2 IV administrations separated by 4 to 5 weeks during the core trial period.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Number analyzed (Observations) | 25
percentage of injected 177Lu-3BP-227
  All cycles: Body: number analyzed (Observations) | 21
  All cycles: Body | 99.7 [99.2 to 100]
  All cycles: Bone marrow: number analyzed (Observations) | 20
  All cycles: Bone marrow | 1.10 [0.560 to 1.98]
  All cycles: Left kidney | 0.247 [0.130 to 0.409]
  All cycles: Right kidney | 0.227 [0.129 to 0.452]
  All cycles: Healthy liver: number analyzed (Observations) | 20
  All cycles: Healthy liver | 1.01 [0.0760 to 1.84]
  All cycles: Spleen: number analyzed (Observations) | 17
  All cycles: Spleen | 0.280 [0.110 to 0.770]

3. Secondary Outcome: Phase 1: Maximal Concentration (Cmax) of 177Lu-3BP-227
Description: The pharmacokinetic (PK) sampling was performed from Day 1 to Day 5 post infusion for each treatment cycle.
Time Frame: Pre-infusion and at the end of infusion, and 5 minutes, 30 minutes, 90 minutes, 4 hours, 24 hours, 48 hours and 72 to 96 hours post infusion in each treatment cycle.
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 1: Time Post Injection to Achieve Cmax of 177Lu-3BP-227
Description: The PK sampling was performed from Day 1 to Day 5 post infusion for each treatment cycle.
Time Frame: as for outcome 3
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Versus Time Curve (AUC) of 177Lu-3BP-227
Description: The PK sampling was performed from Day 1 to Day 5 post infusion for each treatment cycle.
Time Frame: as for outcome 3
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 1: Half-life (t1/2) of 177Lu-3BP-227
Description: The PK sampling was performed from Day 1 to Day 5 post infusion for each treatment cycle.
Time Frame: as for outcome 3
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 1: Number of Participants With Highest Absorbed Dose of 177Lu-3BP-227 to Each Discernible Organ
Description: The absorbed dose to the target lesions and discernible organs (i.e., organs showing uptake) was evaluated by image-based analysis. The organs considered for 177Lu-3BP-227 image-based dosimetry assessment included: healthy liver, total liver, bone marrow, left kidney, right kidney, intestine (large and small), spleen, pancreas, stomach wall, right ovary, left ovary, uterus, right testis, left testis, thymus, right thyroid gland, left thyroid gland, prostate gland and total body. The organ that had the highest absorbed dose of treatment for each participant in each treatment cycle was determined.
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: Dosimetry population included all participants with organ dosimetry data and with no major protocol deviations with an impact on dosimetry analysis. Since the study drug administered to the different groups had the same composition/specific activity, no difference in drug distribution was expected between groups and results were reported combining all groups.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  Cycle 1: Right kidney | 4
  Cycle 1: Left kidney | 3
  Cycle 1: Large intestine | 5
  Cycle 1: Bladder | 2
  Cycle 1: Lymph node | 0
  Cycle 2: number analyzed (Participants) | 11
  Cycle 2: Right kidney | 2
  Cycle 2: Left kidney | 2
  Cycle 2: Large intestine | 4
  Cycle 2: Bladder | 2
  Cycle 2: Lymph node | 1

8. Secondary Outcome: Phase 1: Specific Absorbed Dose to the Target Lesions of 177Lu-3BP-227
Description: The specific absorbed dose to the target lesions was evaluated by image-based analysis. Results for all studied diseases (pancreatic ductal adenocarcinoma and colorectal carcinoma) at all anatomical locations (cervical, intrapelvic, liver, lung, lymph node, and pancreas) for all cycles (Cycle 1 and 2) are reported. The specific absorbed dose (Gray/GBq) was calculated as the absorbed dose to the target lesions (in Gray) divided by the activity of 177Lu-3BP-227 administered (in GBq).
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: Dosimetry population included all participants with organ dosimetry data and with no major protocol deviations with an impact on dosimetry analysis. Since study drug administered to different groups had same composition/specific activity and since the specific absorbed dose is expressed relatively to the administered activity (Gray/Gbq), no difference in specific absorbed dose was expected between groups and results were reported combining all groups.
Measure: Median (Full Range); unit: Gray/GBq
Units Other Than Participants: Lesions
Arm/Group | All Participants
Number analyzed (Participants) | 14
Number analyzed (Lesions) | 47
Gray/GBq | 0.183 [0.0551 to 1.21]

9. Secondary Outcome: Phase 1: Specific Absorbed Dose Per Organ of 177Lu-3BP-227
Description: The specific absorbed dose per organ was evaluated by image-based analysis. The specific absorbed dose (Gray/GBq) was calculated as the absorbed dose to an organ (in Gray) divided by the activity of 177Lu-3BP-227 administered (in GBq).
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: as for outcome 8
Measure: Median (Full Range); unit: Gray/GBq
Units Other Than Participants: Observations of injected 177Lu-3BP-227
Arm/Group | All Participants
Number analyzed (Participants) | 14
Number analyzed (Observations of injected 177Lu-3BP-227) | 25
Gray/GBq
  All cycles: Bone marrow | 0.0636 [0.0346 to 0.0943]
  All cycles: Healthy liver | 0.0515 [0.0263 to 0.0811]
  All cycles: Left kidney | 0.255 [0.102 to 1.05]
  All cycles: Right kidney | 0.242 [0.118 to 0.943]

10. Secondary Outcome: Phase 1: Cumulative Absorbed Organ Doses of 177Lu-3BP-227
Description: The cumulative absorbed dose to the discernible organs (i.e., organs showing uptake) was evaluated by image-based analysis.
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: Dosimetry population included all participants with organ dosimetry data and with no major protocol deviations with an impact on dosimetry analysis. Cumulative absorbed doses on Cycles 1 and 2 are only presented for participants who have performed the 2 cycles.
Measure: Median (Full Range); unit: Gray
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 1
Gray
  Cycle 2: Bone marrow | 0.326 [0.326 to 0.326] | 0.604 [0.304 to 0.645] | 0.680 [0.391 to 0.837] | 0.820 [0.628 to 1.11] | 0.694 [0.694 to 0.694]
  Cycle 2: Healthy liver | 0.254 [0.254 to 0.254] | 0.353 [0.271 to 0.415] | 0.530 [0.428 to 0.637] | 0.714 [0.469 to 0.927] | 0.571 [0.571 to 0.571]
  Cycle 2: Left kidney | 2.17 [2.17 to 2.17] | 4.19 [1.38 to 6.21] | 3.33 [1.90 to 5.12] | 3.44 [1.90 to 3.48] | 2.95 [2.95 to 2.95]
  Cycle 2: Right kidney | 2.38 [2.38 to 2.38] | 3.39 [1.53 to 5.51] | 2.97 [2.14 to 5.74] | 3.01 [2.00 to 4.67] | 2.92 [2.92 to 2.92]

11. Secondary Outcome: Phase 1: Cmax of 3BP-227
Description: The PK sampling was performed from Day 1 to Day 3 post infusion of 177Lu-3BP-227 in Cycle 1.
Time Frame: Pre-infusion and at the end of infusion, and 5 minutes, 30 minutes, 90 minutes, 4 hours, 6 hours, 8 hours, 24 hours and 48 hours post infusion of 177Lu-3BP-227 in Cycle 1.
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase 1: AUC of 3BP-227
Description: The PK sampling was performed from Day 1 to Day 3 post infusion of 177Lu-3BP-227 in Cycle 1.
Time Frame: as for outcome 11
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 1: t1/2 of 3BP-227
Description: The PK sampling was performed from Day 1 to Day 3 post infusion of 177Lu-3BP-227 in Cycle 1.
Time Frame: as for outcome 11
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 1: Clearance of 3BP-227
Description: The PK sampling was performed from Day 1 to Day 3 post infusion of 177Lu-3BP-227 in Cycle 1.
Time Frame: as for outcome 11
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 1: Volume of Distribution of 3BP-227
Description: The PK sampling was performed from Day 1 to Day 3 post infusion of 177Lu-3BP-227 in Cycle 1.
Time Frame: as for outcome 11
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase 1: Cumulative Amount of Unchanged 3BP-227 Excreted Into the Urine
Description: The PK sampling was performed from Day 1 to Day 3 post infusion of 177Lu-3BP-227 in Cycle 1.
Time Frame: as for outcome 11
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase 1: Renal Clearance of 3BP-227 From Plasma
Description: The PK sampling was performed from Day 1 to Day 3 post infusion of 177Lu-3BP-227 in Cycle 1.
Time Frame: as for outcome 11
Population: Due to the early termination of the study, the PK analysis data was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

18. Secondary Outcome: Phase 1: Number of Participants With Objective Response Rate (ORR)
Description: The ORR was defined as number of participants with a best overall response (BOR) characterized as either a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) relative to the total number of evaluable participants.
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: Primary Pharmacodynamic population (for tumor response) included all participants who received at least 2 therapeutic doses of 177Lu-3BP-227 and reached the end of Cycle 2 or EOCT visit with available post-baseline tumor assessment based on RECIST 1.1 and with no major protocol deviations with an impact on the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 1
Participants | 0 | 1 | 0 | 0 | 0

19. Secondary Outcome: Phase 1: Number of Participants With Disease Control Rate (DCR)
Description: The DCR was defined as number of participants with a BOR characterized as CR, PR or stable disease according to RECIST 1.1 relative to the total number of evaluable participants.
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 1
Participants | 0 | 1 | 0 | 0 | 0

20. Secondary Outcome: Phase 1: Progression-Free Survival (PFS)
Description: The PFS was defined as the time from date of first study medication administration until progression, according to RECIST 1.1.
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: Due to the early termination of the study, survival analysis on PFS was not collected.
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Phase 1: Overall Survival (OS)
Description: The OS was defined from first study medication administration until death, according to RECIST 1.1.
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: Due to the early termination of the study, survival analysis on OS was not collected.
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Phase 1: Metabolic Tumor Response Using Positron Emission Tomography (PET) Response Criteria In Solid Tumors (PERCIST) Version 1.0 or Practical PERCIST
Description: Tumor response assessments were planned to perform by the site investigator (local) for the phase 1 and dose escalation part and by independent reader (central) for the phase 2. All fluorine-18 fluorodeoxyglucose-PET images were used for the metabolic tumor response assessments as described in PERCIST version 1.0 by the Investigator and/or independent readers.
Time Frame: From the start of the first study medication (Day 1) up to EOCT, maximum of 16 weeks.
Population: Due to the early termination of the study, metabolic tumor response was not collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

23. Secondary Outcome: Phase 1: Tumor Marker Levels in Serum - Cancer Antigen 19-9
Description: Changes in tumor markers in serum relevant and specific to the underlying tumor disease was determined.
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, EOCT (maximum of 16 weeks) and early withdrawal
Population: Pharmacodynamic population included all participants who received at least 1 therapeutic dose and with available post-baseline pharmacodynamics/efficacy data.
Measure: Mean (Standard Deviation); unit: international units/milliliter
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Number analyzed (Participants) | 2 | 3 | 5 | 3 | 1
international units/milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 1 | 5 | 2 | 1
  Cycle 1 Day 1 | 50019.00 (70683.81) | 13.00 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 20939.54 (46482.66) | 1455.50 (78.49) | 314.70 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed.
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 3 | 3 | 3 | 1
  Cycle 2 Day 1 | 66.00 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 456.33 (753.23) | 277.90 (239.71) | 18420.33 (27442.99) | 490.50 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed.
  EOCT: number analyzed (Participants) | 1 | 2 | 1 | 1 | 1
  EOCT | 112.00 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 928.00 (1294.01) | 1166.90 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 3532.00 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 629.90 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed.
  Early Withdrawal: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0
  Early Withdrawal |  |  | 64.90 (86.41) | 8398.00 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. |

24. Secondary Outcome: Phase 1: Tumor Marker Levels in Serum - Carcinoembryonic Antigen
Description: Changes in tumor markers in serum relevant and specific to the underlying tumor disease was determined.
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, EOCT (maximum of 16 weeks) and early withdrawal
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: microgram per liter
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
Number analyzed (Participants) | 2 | 3 | 5 | 3 | 1
microgram per liter
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 1 | 5 | 2 | 1
  Cycle 1 Day 1 | 857.95 (1209.22) | 117.40 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 112.38 (94.41) | 6.65 (7.14) | 3.50 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed.
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 3 | 3 | 3 | 1
  Cycle 2 Day 1 | 3.20 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 37.93 (41.01) | 210.97 (213.86) | 47.87 (62.85) | 4.60 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed.
  EOCT: number analyzed (Participants) | 1 | 2 | 1 | 1 | 1
  EOCT | 4.30 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 75.50 (47.09) | 321.20 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 184.00 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. | 5.10 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed.
  Early Withdrawal: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0
  Early Withdrawal |  |  | 53.75 (23.83) | 29.60 (NA) — Standard deviation cannot be calculated when only 1 participant analyzed. |

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported for participants who received the therapeutic dose of 177Lu-32P-227 during the core trial (Cycle 1 Day 1 up to EOCT); maximum of 16 weeks.
Description: Safety population contained all participants who received at least 1 dose of study medication.
Arm/Group | Cohort 1: 177Lu-3BP-227 2.5 GBq | Cohort 2: 177Lu-3BP-227 4.0 GBq | Cohort 3: 177Lu-3BP-227 5.5 GBq | Cohort 4: 177Lu-3BP-227 6.5 GBq | Cohort 5: 177Lu-3BP-227 7.5 GBq
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/3 | 2/5 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/3 | 5/5 | 3/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 5/5 | 3/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 177Lu-3BP-227 2.5 GBq (N=2) | Cohort 2: 177Lu-3BP-227 4.0 GBq (N=3) | Cohort 3: 177Lu-3BP-227 5.5 GBq (N=5) | Cohort 4: 177Lu-3BP-227 6.5 GBq (N=3) | Cohort 5: 177Lu-3BP-227 7.5 GBq (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 177Lu-3BP-227 2.5 GBq (N=2) | Cohort 2: 177Lu-3BP-227 4.0 GBq (N=3) | Cohort 3: 177Lu-3BP-227 5.5 GBq (N=5) | Cohort 4: 177Lu-3BP-227 6.5 GBq (N=3) | Cohort 5: 177Lu-3BP-227 7.5 GBq (N=1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 2 (7) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (8) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 3 (6) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Illusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Product prescribing error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The sponsor terminated the study early and phase 1 dose expansion and phase 2 were not started. The decision to terminate the study was not due to any safety or tolerability concern, or any event associated with the use of 177Lu-3BP-227.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT03525392/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT03525392/SAP_001.pdf